CLINICAL TRIAL: NCT07312396
Title: An Exploratory Clinical Study on the Protective Effect of Cycling on the Ankle Joint in Gout
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhu Xiaoxia (Other)
Responsible Party: Sponsor-Investigator, Zhu Xiaoxia, Associate Chief Physician, Huashan Hospital
Organization: Huashan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KY2025-872
Record Dates: First submitted 2025-09-14; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Gout Arthritis; Cycling; Physical Activity
MeSH Terms: conditions — Arthritis, Gouty; Motor Activity | interventions — Jogging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator)
  Interventions: Drug: Urate-lowering therapy (ULT); Behavioral: Jogging
- Experimental Group (Experimental)
  Interventions: Drug: Urate-lowering therapy (ULT); Behavioral: Cycling

INTERVENTIONS:
Drug: Urate-lowering therapy (ULT) — The treatment with uric acid-lowering drugs remained the same as the standard uric acid-lowering treatment plan at the time of enrollment
Behavioral: Jogging — Participants in the study could exercise on the treadmills in the fitness center or jog outdoors, but both needed to reach a moderate intensity. Each total exercise session lasts between 45 and 60 minutes (including 5 to 10 minutes of warm-up time, no less than 20 minutes of exercise time reaching 65% to 75% of the maximum heart rate, and 10 to 15 minutes of cool-down exercise/muscle stretching time).
  Arms: Control Group
Behavioral: Cycling — Participants in the study could use the cycling equipment at the fitness center for exercise or do cycling outdoors, but both needed to reach a moderate intensity. Each total exercise session lasts between 45 and 60 minutes (including 5 to 10 minutes of warm-up time, no less than 20 minutes of exercise time reaching 65% to 75% of the maximum heart rate, and 10 to 15 minutes of cool-down exercise/muscle stretching time).
  Arms: Experimental Group

SUMMARY:
This study divided the enrolled gout patients into a jogging group and a cycling group to investigate 1）the effectiveness of cycling intervention in reducing the recurrence risk of gouty ankle arthritis compared with jogging. 2) To clarify the influence of different exercise patterns on the ultrasonic manifestations of gouty ankle arthritis; 3) Clarify the impact of different exercise methods on the blood uric acid levels of gout patients;

ELIGIBILITY:
Inclusion Criteria:

* meets the diagnostic criteria for gout of the American College of Rheumatology (ACR) and the European League Against Rheumatism (EULAR) in 2015
* There have been two histories of gout attacks on either side of the ankle joint in the past six months
* Ultrasound examination within the past 6 months indicated that either ankle joint had characteristic ultrasound manifestations (double-track sign, and/or hyperechoic aggregates, and/or tophi, and/or bone destruction)
* Those who have had an interval of at least 4 weeks since the most recent acute gout attack
* If the patient is undergoing uric acid-lowering drug treatment, the drug dosage must remain stable for more than 4 weeks. During the study period, the uric acid-lowering drug regimen or dosage will not be adjusted
* For women who have the potential to become pregnant, a pregnancy test must be negative, they must not be in the lactation period, and it must be confirmed that they are receiving contraception approved by the researcher and agree to maintain this contraceptive measure throughout the study process
* Those who were informed of this study and signed the informed consent form

Exclusion Criteria:

* Those who have received intra-articular injections of corticosteroids during an attack within the past three months; Those who have taken colchicine, NSAIDs, glucocorticoids in the past two weeks, or those who need to maintain anti-inflammatory drug treatment for a long time during the follow-up period
* Joint trauma or other types of arthritis
* There is a history of joint prosthesis or joint surgery
* Those who have had acute gout attacks within 4 weeks
* Patients with secondary gout caused by kidney diseases, blood disorders, or taking certain medications, radiotherapy and chemotherapy for tumors, etc
* Those with severe and unstable cardiovascular and cerebrovascular diseases (such as unstable angina pectoris, coronary angiogenesis, cerebral angiogenesis, transient ischemic attack, congestive heart failure, etc.) and other diseases that researchers have determined to be acute and difficult to control

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
The frequency of gout attacks | From enrollment to the end of treatment at 24 weeks

SECONDARY OUTCOMES:
blood uric acid | From enrollment to the end of treatment at 24 weeks
Gouty arthritis joint pain score | From enrollment to the end of treatment at 24 weeks
Ankle joint magnetic resonance | From enrollment to the end of treatment at 24 weeks
Ankle joint ultrasound | From enrollment to the end of treatment at 24 weeks

OTHER OUTCOMES:
Incidence and severity of adverse events/serious adverse events | From enrollment to the end of treatment at 24 weeks

IPD SHARING:
Plan to Share IPD: Yes